CLINICAL TRIAL: NCT06559878
Title: Hepatic Mitochondrial Metabolism in Fatty Liver Disease in Humans
Acronym: ALPHA
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Panu Luukkonen, MD, PhD, Helsinki University Central Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HUS/8748/2023
Record Dates: First submitted 2024-08-12; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Non-alcoholic Fatty Liver Disease NAFLD
Keywords: Hepatic mitochondrial dysfunction; MAFLD; Non-alcoholic Fatty Liver Disease NAFLD; 13C-α-Ketoisocaproic Acid Breath Test
MeSH Terms: interventions — Ethanol; Fat Emulsions, Intravenous; Saline Solution

STUDY DESIGN:
Intervention Model Description: The study protocol includes five clinical visits. At first visit, an informed consent will be obtained, followed by assessment of inclusion/exclusion criteria. Participants fulfilling the criteria will be enrolled in the study. At second visit, magnetic resonance studies will be performed to quantify liver fat content. Visits 3-5 consist of metabolic studies using the 13C-ketoisocaproate breath test and, in a random order, infusions of either a) saline alone, b) saline, a lipid emulsion and heparin or c) saline and ethanol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- The order of metabolic visits: 1.Normal saline, 2.Lipid emulsion, 3.Ethanol (Experimental)
  Interventions: Diagnostic Test: 13C-α-Ketoisocaproic Acid Breath Test; Dietary Supplement: Ethanol; Dietary Supplement: Lipid Emulsion; Other: Normal Saline
- The order of metabolic visits: 1. Normal saline, 2. Ethanol, 3. Lipid emulsion (Experimental)
  Interventions: Diagnostic Test: 13C-α-Ketoisocaproic Acid Breath Test; Dietary Supplement: Ethanol; Dietary Supplement: Lipid Emulsion; Other: Normal Saline
- The order of metabolic visits: 1.Lipid emulsion, 2.Normal saline, 3.Ethanol (Experimental)
  Interventions: Diagnostic Test: 13C-α-Ketoisocaproic Acid Breath Test; Dietary Supplement: Ethanol; Dietary Supplement: Lipid Emulsion; Other: Normal Saline
- The order of metabolic visits: 1.Lipid emulsion, 2.Ethanol, 3.Normal saline (Experimental)
  Interventions: Diagnostic Test: 13C-α-Ketoisocaproic Acid Breath Test; Dietary Supplement: Ethanol; Dietary Supplement: Lipid Emulsion; Other: Normal Saline
- The order of metabolic visits: 1. Ethanol, 2. Normal saline, 3. Lipid emulsion (Experimental)
  Interventions: Diagnostic Test: 13C-α-Ketoisocaproic Acid Breath Test; Dietary Supplement: Ethanol; Dietary Supplement: Lipid Emulsion; Other: Normal Saline
- The order of metabolic visits: 1. Ethanol, 2. Lipid emulsion, 3. Normal saline (Experimental)
  Interventions: Diagnostic Test: 13C-α-Ketoisocaproic Acid Breath Test; Dietary Supplement: Ethanol; Dietary Supplement: Lipid Emulsion; Other: Normal Saline

INTERVENTIONS:
Diagnostic Test: 13C-α-Ketoisocaproic Acid Breath Test — 13C-α-Ketoisocaproic acid with L-Leucine soluted in citric acid drink. The solution is administered orally during metabolic visits (3.-5.).
Dietary Supplement: Ethanol — 6% ethanol soluted in normal saline is given intravenously during one metabolic visit.
  Other Names: Alcohol
Dietary Supplement: Lipid Emulsion — Lipid emulsion, heparin and normal saline are given intravenously during one metabolic visit.
Other: Normal Saline — Normal saline is given intravenously during one metabolic visit.

SUMMARY:
The goal of this clinical trial is to investigate in healthy volunteers the mechanisms by which ethanol and lipids, the two key risk factors of steatotic liver disease (SLD), affect liver mitochondrial metabolism.

The main question it aims to answer is:

• Does acute administration of ethanol and lipids increase hepatic mitochondrial reductive stress as determined by orally ingested stable isotope tracer 13C-alpha-ketoisocaproate and by plasma beta-hydroxybutyrate to acetoacetate ratio (b-OHB/AcAc) in humans?

DETAILED DESCRIPTION:
In this study we investigate the effects of ethanol and lipids on hepatic mitochondrial metabolism in healthy volunteers.

At first visit, an informed consent will be obtained, followed by assessment of inclusion/exclusion criteria. Participants fulfilling the criteria will be enrolled in the study. Body composition will be determined with bioelectrical impedance.

At second visit hepatic lipid content will be measured with magnetic resonance spectroscopy.

Participants will be given in random order on three separate visits (3-5):

* Intravenous infusion of ethanol and normal saline (breath alcohol content target and upper limit corresponding to 0.6 per mil in blood)
* Intravenous infusions of lipid emulsion, heparin and normal saline
* Intravenous infusion of normal saline

On study visits participant will drink a tracer dose of 13C-alpha-ketoisocaproate and L-Leucine. Breath samples are collected at different time points for determination of 13C enrichment of CO2. Furthermore "arterialized" blood samples are taken during study visits to obtain beta-hydroxybutyrate to acetoacetate ratios (b-OHB/AcAc) at different timepoints.

Whole-body oxidation of lipids, carbohydrates and protein will be determined using indirect calorimetry.

ELIGIBILITY:
1. Participants must be able to communicate meaningfully with the investigator and must be legally competent to provide written informed consent.
2. Subject must be likely to be available to complete all protocol-required study visits or procedures, to the best of the subject's and investigator's knowledge.
3. Age range from 18-75 years.
4. No known hypersensitivity to egg, soy, or peanut protein, or to any of the substances of Intralipid 20%, or to any other substance to be administered during the study.
5. No severe hyperlipidemia or hemophagocytotic syndrome as judged by history and physical examination and standard laboratory tests.
6. No other liver disease except for SLD.
7. No advanced liver disease as judged by history and physical examination and standard laboratory tests.
8. No claustrophobia or metal implants to allow magnetic resonance studies.
9. No pregnancy or lactation in women.
10. No known or anticipated difficulties in cannulation of peripheral veins.
11. No history or evidence of any other clinically significant disorder, condition or disease other than those outlined above that, in the opinion of the investigator may compromise the ability of the subject to give written informed consent, would pose a risk to subject safety, or interfere with the study evaluation, procedures or completion.
12. No drinking problem based on AUDIT questionnaire.
13. No use of medications interacting with alcohol.
14. No history of heparin induced thrombosytopenia (HIT) or bleeding tendency.
15. No current use of warfarin, direct anticoagulants, or thrombocyte inhibitors.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in arterialized plasma b-OHB to AcAc ratio | From baseline to the end of treatment at 240 minutes
  Arterialized plasma b-OHB and AcAc concentrations
Breath 13CO2 enrichment after ingesting 13C-alpha-ketoisocaproate | From baseline to the end of treatment at 330 minutes.
  Measured as area under the curve

OTHER OUTCOMES:
Plasma metabolomics | From baseline until the end of treatment at 240 minutes.
  Arterialized plasma analyzed by nuclear magnetic resonance and mass spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: Panu Luukkonen, MD, PhD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Helsinki Central University Hospital, Helsinki, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: No
Due to European Union GDPR regulations.